CLINICAL TRIAL: NCT07153835
Title: Evaluation of Efficacy and Safety of Paliperidone Among People With Schizophrenia in Bangladesh
Brief Title: Efficacy and Safety of Paliperidone in Schizophrenia - Bangladesh Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sher-E-Bangla Medical College (Other)
Collaborators: ACI Pharmaceuticals (Unknown); US-Bangla Medical College Hospital (Unknown); Dr. M M Jalal Uddin (Unknown); Dr.Ahsan Aziz Sarkar (Unknown)
Responsible Party: Principal Investigator, Mohammad Tariqul Alam, Professor, Sher-E-Bangla Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB/USBMC/2025/001
Record Dates: First submitted 2025-08-16; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Extended-Release Paliperidone; Second-Generation Antipsychotics; PANSS; GASS; WHOQOL-BREF; Quasi-Experimental Study; Efficacy; Safety
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-level, multicenter, prospective, quasi-experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paliperidone Extended-Release Treatment Arm (Experimental): Participants in this arm will receive paliperidone extended-release (ER) tablets at a flexible daily dose of 6-12 mg, as determined by the treating psychiatrist based on clinical judgment. The treatment will continue for 12 weeks, with clinical assessments at baseline, 6 weeks, and 12 weeks to evaluate efficacy, safety, and quality of life.
  Interventions: Drug: Paliperidone extended-release (ER)

INTERVENTIONS:
Drug: Paliperidone extended-release (ER) — Paliperidone extended-release (ER) tablets will be administered orally once daily at flexible doses ranging from 6 mg to 12 mg, based on the clinical judgment of the treating psychiatrist. The treatment duration is 12 weeks. Dose adjustments may be made throughout the study period depending on patient response and tolerability.

SUMMARY:
This is a single-arm, open-label, multicenter, prospective quasi-experimental study evaluating the efficacy and safety of extended-release paliperidone in adults with schizophrenia in Bangladesh. The study will assess psychotic symptom improvement using the PANSS scale, monitor side effects using GASS, and evaluate quality of life via WHOQOL-BREF.

DETAILED DESCRIPTION:
Despite global evidence supporting the effectiveness of paliperidone, there is limited data from low- and middle-income countries such as Bangladesh. This study addresses this evidence gap by assessing the efficacy and safety of paliperidone ER in a real-world, multi-site setting. The primary endpoint is the change in PANSS score after 12 weeks of treatment. Secondary outcomes include side-effect profile, safety assessments, and quality of life. A total of 505 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years
* Diagnosed with schizophrenia according to DSM-5 criteria
* At least 3 months since the initial diagnosis of schizophrenia
* Either antipsychotic-naïve or previously treated with one antipsychotic but requiring a change due to non-response, poor response, or intolerable side effects. (If previously treated, a washout period of 7 days before study medication initiation)
* PANSS (Positive and Negative Syndrome Scale) total score ≥70
* Clinically stable for at least 2 weeks before enrollment

Exclusion Criteria:

* History of being diagnosed with treatment-resistant schizophrenia
* Comorbid severe medical or neurological conditions
* Pregnant or lactating women
* Previous known hypersensitivity to paliperidone or risperidone
* Use of long-acting injectable antipsychotics within the last 3 months
* Current diagnosis of substance related disorder or substance misuse in the previous month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 505 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in PANSS total score from baseline to 12 weeks | Baseline, Week 6, Week 12
  The Positive and Negative Syndrome Scale (PANSS) will be used to assess the severity of schizophrenia symptoms. The total score ranges from 30 to 210, with higher scores indicating more severe symptoms. The primary outcome is the change in total PANSS score from baseline to week 12 following treatment with paliperidone extended-release.

SECONDARY OUTCOMES:
Assessment of Side Effects Using GASS Score | Baseline, Week 6, and Week 12
  The Glasgow Antipsychotic Side-Effect Scale (GASS) will be used to assess self-reported side effects of paliperidone. For participants who are not literate or have difficulty completing the form independently, a trained psychiatrist will administer the scale in an interview format.
Changes in Quality of Life Measured by WHOQOL-BREF | Baseline and Week 12
  The WHO Quality of Life-BREF (WHOQOL-BREF) will be used to assess quality of life across four domains: physical health, psychological health, social relationships, and environment. For participants who are not literate, the questionnaire will be administered by a trained psychiatrist through structured interviews.

OTHER OUTCOMES:
Changes in Laboratory Parameters and ECG | Baseline and Week 12
  Safety will be assessed through laboratory investigations including complete blood count, liver and renal function tests, fasting glucose, and lipid profile, as well as 12-lead ECG. Abnormal values or clinically significant changes from baseline will be recorded.
Change in Body Mass Index (BMI) | Baseline, Week 6, and Week 12
  BMI will be calculated as weight (kg) divided by height squared (m²). Height will be measured once at Baseline (without shoes, using a stadiometer) and used for all BMI calculations. Weight will be measured at each visit on a calibrated digital scale with participants in light clothing and no shoes. The reported outcome will be BMI (kg/m²) at each time point and the change from Baseline. Weight and height are collected only to compute BMI and will not be reported as separate outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. M M Jalal Uddin Co-invetigator, MBBS,FCPS (Psychiatry), MPH, Study Director — National Institute of Neurosciences and Hospital
Locations (1):
- Sher-E-Bangla Medical College Hospital, Barishal, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may not be shared publicly, as the decision to share lies with the trial sponsor, ACI Pharmaceuticals.